CLINICAL TRIAL: NCT04771078
Title: Expanded Access Protocol (EAP) for Patients Receiving Idecabtagene Vicleucel That is Nonconforming for Commercial Release
Brief Title: Expanded Access Protocol (EAP) for Participants Receiving Idecabtagene Vicleucel That is Nonconforming for Commercial Release
Status: Available | Type: Expanded Access
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: BB2121-EAP-001; U1111-1263-0642 (Registry Identifier: WHO)
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: BB2121; Multiple Myeloma; Expanded Access; idecabtagene vicleucel; nonconforming; CAR T; EAP; Pre-Approval Access
MeSH Terms: conditions — Multiple Myeloma | interventions — idecabtagene vicleucel

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: Nonconforming idecabtagene vicleucel — Nonconforming idecabtagene vicleucel is to be administered to participants after lymphodepleting chemotherapy
  Other Names: BB2121

SUMMARY:
This study is designed to evaluate the safety and efficacy of nonconforming idecabtagene vicleucel (ide-cel) in participants with multiple myeloma per the approved prescribing information. This is an expanded access protocol (EAP) to be conducted at Risk Evaluation and Mitigation Strategies (REMS) qualified sites approved for commercial administration of idecabtagene vicleucel and where the EAP is authorized to be conducted for use of nonconforming idecabtagene vicleucel.

Non-conforming idecabtagene vicluecel is idecabtagene vicleucel that does not meet commercial release specifications but may be acceptable for use as an investigational product in the Expanded Access Protocol setting.

ELIGIBILITY:
Inclusion Criteria:

* Had a participant-specific batch of Idecabtagene vicleucel (ide-cel) manufactured intended for commercial treatment; however, the final manufactured product was nonconforming and did not meet commercial release criteria
* Remanufacturing is deemed not feasible or clinically inappropriate per assessment of the treating physician in discussion with the participant
* Clinically stable

Exclusion Criteria:

* Has a hypersensitivity to the active substance or to any of the excipients
* No experience of a significant worsening in clinical status that would, in the opinion of the treating physician, either increase the risk of Adverse Events associated with lymphodepleting chemotherapy, or exclude them from treatment with nonconforming Idecabtagene vicleucel (ide-cel)
* Has any condition and/or laboratory abnormality that places the participant at unacceptable risk if he/she were to participate in the Expanded Access Protocol based on the Investigator's judgement

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html